CLINICAL TRIAL: NCT02655575
Title: Assessment and Treatment of Patients With Long-term Dizziness in Primary Care
Acronym: LODIP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bergen University College (Other)
Collaborators: University of Bergen (Other); Norwegian Fund for Postgraduate Training in Physiotherapy (Other); University of Southern Denmark (Other); Duke University (Other); Haukeland University Hospital (Other)
Responsible Party: Principal Investigator, Liv Heide Magnussen, Associated Professor, ph.d., Bergen University College
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2014/921
Record Dates: First submitted 2015-11-10; First posted 2016-01-14 (Estimated); Last update posted 2025-02-05 (Actual); Status verified 2025-02

CONDITIONS: Dizziness; Vertigo; Vestibular Neuritis
Keywords: dizziness; cognitive therapy; primary care; vestibular rehabilitation; chronic
MeSH Terms: conditions — Dizziness; Vertigo; Vestibular Neuronitis; Bronchiolitis Obliterans Syndrome | interventions — Crisis Intervention; Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- BI + VR + CBT (Experimental): Brief Intervention (BI) consists of an individual clinical examination, education/information and advice about being active Vestibular Rehabilitation (VR) includes active exercises that provokes dizziness, Balance exercises and body awareness exercises in a group format.
  Cognitive Behavioral Therapy (CBT) includes conversation and reflection about factors that may be a barrier to Activity and participation
  Interventions: Behavioral: BI + VR + CBT; Behavioral: BI + phone calls
- BI + phone calls (Active Comparator): Brief Intervention (BI) consists of an individual clinical examination, education/information and advice about being active Phone Calls as follow-up at week 2 and 6 to reassure
  Interventions: Behavioral: BI + VR + CBT; Behavioral: BI + phone calls

INTERVENTIONS:
Behavioral: BI + VR + CBT — Brief intervention (information and advice) + group-based vestibular rehabilitation combined with cognitive behavioral therapy
  Other Names: Brief intervention (BI); Vestibular rehabilitation (VR); Cognitive behavioral therapy (CBT)
Behavioral: BI + phone calls — Brief intervention (information and advice). Patients are followed-up by phone calls
  Other Names: Brief intervention (BI)

SUMMARY:
Brief Summary:

The purpose of the present study is to examine the effects of a Group based intervention consisting of vestibular rehabilitation (VR) combined with cognitive behavioral therapy (CBT) in patients with long--lasting vestibular dizziness. The study also aims to describe sociodemographic, physical and psychological characteristics in the patients, and to examine prognostic factors related to functional status and disability following participation in the intervention.

Prior to the RCT, a feasibility study will be conducted to examine the feasibility of the study protocol.

DETAILED DESCRIPTION:
Dizziness is a common complaint. International studies show a prevalence of balance/dizziness problems in 10-30% in the population, and in Norway it is reported that 11 % of the population have symptoms of dizziness and/or imbalance during the last three months. Peripheral vestibular disorders are the most common cause of dizziness presenting in primary care. Most people recover within a few weeks , but it is assumed that about 30% of the patients do not recover fully from an acute peripheral vestibular disorder and develop long-lasting dizziness, often with secondary musculoskeletal pain and anxiety, making it a multifactorial syndrome. It is unknown if these secondary complaints are issues that maintain or exacerbates the dizziness, or if a high level of musculoskeletal and psychological problems may predict future disability.There is a general consensus that exercises labeled as Vestibular Rehabilitation (VR) is the most effective treatment for vestibular dysfunction. VR exercises involve eye, head and body movements aiming to provoke dizziness, which is a prerequisite for adaptation and recovery. However, not all patients will recover from VR, and therefore increased attention toward the psychological aspects, targeting how patients think about the dizziness has been addressed. Cognitive behavioral therapy (CBT) alone or in addition to VR seems to have limited effect. This present study aims to combine an existing group treatment targeting body awareness and VR with CBT in order to address both the movement provoked dizziness and secondary complaints that patients with long-term dizziness often present with.

Prior to conducting the RCT the feasibility of recruitment procedures, test procedures and the interventions (CBT-VR and BI) will be examined in a feasibility study. The study is judged as feasible if the participants could complete the testing and adhere to the treatment protocols, of they found the intervention appropriate for their complaints, and if the primary outcomes improved following the intervention. Eight participants were planned for the study.

ELIGIBILITY:
Inclusion Criteria:

* The dizziness is provoked or aggravated by head movements, more than 3 months duration og symptoms, the dizziness started acute, understand Norwegian

Exclusion Criteria:

* Dizziness no longer a problem, other known reasons, than vestibular, for the dizziness (neurological, psychological, or cancer), fluctuating vestibular disease (e.g, ménières disease), scheduled for treatment of/ have had treatment for benign paroxysmal positional vertigo within one month,conditions where fast head movements are contraindicated (e.g. osteoporosis of the neck, whiplash associated injuries), participated in group therapy for dizziness within the past year, unable to attend test and treatment locations

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2015-10 (Actual); Primary Completion 2022-05-31 (Actual); Study Completion 2022-05-31 (Actual)

PRIMARY OUTCOMES:
Dizziness Handicap Inventory (DHI) | 3 min
6 m walking test preferred velocity | 5 min
  6 meter walking distance (preferred velocity) measured in Seconds. Mean of two trials

SECONDARY OUTCOMES:
Vertigo symptom scale (VSS-SF) | 3 min
Patient Specific Functional Scale (PSFS) | 3 min
Subjective Health Complaints (SHC) | 3 min
Body Sensation Questionnaire (BSQ) | 3 min
Mobility Index (MI-A) | 3 min
Panic Attack Scale (PAS) | 3 min
EQ-5D-5L | 2 min
Hospital Anxiety and Depression Scale (HADS) | 3 min
Global Muscle Examination (GME) - flexibility | 6 min
Patient Global Impression of Change | 1 min
Dynamic Visual Aquity Test (DVA) | 2 min
Hand Grip test | 2 min
6 m walking test (as fast as possible), mean of two test trials | 3 min
  walk 6 meter as fast as possible
Dual task waling test, 6 m | 3 min
  6 meter walking test, optional speed, while doing a cognitive task
Perceived dizziness before and after 1 min head movements | 2 min
The Modified Clinical Test for Sensory Interaction and Balance (mCTSIB) 192 (mCTSIB) test | 4 min
Chalder Fatigue Scale (CFS) | 1 min
Limits of stability (LOS) | 2

CONTACTS AND LOCATIONS:
Overall Officials: Gro AF Flaten, ph.d., Study Director — Bergen University College
Locations (1):
- Bergen University College, Bergen, Norway

REFERENCES:
- [Derived] Kristiansen L, Magnussen LH, Wilhelmsen KT, Maeland S, Nordahl SHG, Clendaniel R, Hovland A, Juul-Kristensen B. Efficacy of intergrating vestibular rehabilitation and cognitive behaviour therapy in persons with persistent dizziness in primary care- a study protocol for a randomised controlled trial. Trials. 2019 Oct 7;20(1):575. doi: 10.1186/s13063-019-3660-5. PMID 31590692
- [Derived] Kristiansen L, Magnussen LH, Juul-Kristensen B, Maeland S, Nordahl SHG, Hovland A, Sjobo T, Wilhelmsen KT. Feasibility of integrating vestibular rehabilitation and cognitive behaviour therapy for people with persistent dizziness. Pilot Feasibility Stud. 2019 May 20;5:69. doi: 10.1186/s40814-019-0452-3. eCollection 2019. PMID 31139431

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-03-22): https://cdn.clinicaltrials.gov/large-docs/75/NCT02655575/Prot_SAP_000.pdf